CLINICAL TRIAL: NCT06073769
Title: Onureg® (Oral Azacitidine) Post-Marketing Surveillance in Korean Patients With Acute Myeloid Leukemia
Brief Title: A Post-Marketing Surveillance Study to Assess the Safety of Oral Azacitidine Maintenance Therapy in Korean Patients With Acute Myeloid Leukemia
Status: Recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA055-007
Record Dates: First submitted 2023-10-03; First posted 2023-10-10 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants receiving oral azacitidine maintenance therapy
  Interventions: Drug: Oral azacitidine

INTERVENTIONS:
Drug: Oral azacitidine — Maintenance therapy according to the approved label

SUMMARY:
The purpose of this observational study is to assess the real-world safety of maintenance therapy with oral azacitidine in Korean participants with acute myeloid leukemia (AML) who achieved first complete remission (CR) or complete remission with incomplete blood count recovery (CRi) following induction chemotherapy with or without consolidation therapy, and who are not eligible for hematopoietic stem cell transplantation (HSCT).

ELIGIBILITY:
Inclusion Criteria:

* Adult participants 19 years of age or older
* Participants who receive oral azacitidine according to the approved label
* For the first 2 years after marketing authorization, all participants who have received or are receiving oral azacitidine will also be registered
* Participants who sign the informed consent form

Exclusion Criteria:

* Participants who are prescribed oral azacitidine for therapeutic indications not approved in Korea
* Participants for whom oral azacitidine is contraindicated per the Korean prescribing information approved by ministry of food and drug safety

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults in Korea with acute myeloid leukemia receiving maintenance therapy with oral azacitidine who achieved first complete remission (CR) or complete remission with incomplete blood count recovery (CRi) following induction chemotherapy with or without consolidation therapy, and who are not eligible for hematopoietic stem cell transplantation (HSCT).
Sampling Method: Non-Probability Sample
Enrollment: 154 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AES) | Up to 12 months
  The type, frequency, seriousness and severity of adverse events (AEs), and relationship of AEs to oral azacitidine

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- South Korea (2):
  - Local Institution - 0001, Seoul
  - Novotech Laboratory Korea Co., Ltd., Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety